CLINICAL TRIAL: NCT02323893
Title: Study of the Kinetics, Dosimetry and Safety of [18F]F-AraG, a Positron Emission Tomography Tracer for Imaging the Activation of the Immune System in Healthy Humans
Brief Title: Study of Kinetics, Dosimetry & Safety of [18F]F-AraG, a Positron Emission Tomography Imaging Tracer in Healthy Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 261201300063
Record Dates: First submitted 2014-12-16; First posted 2014-12-24 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Cancer
Keywords: Positron Emission Tomography; Cancer Immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-FAraG (Experimental): A single dose intravenous injection of 18F-FAraG followed by PET scanning.
  Interventions: Drug: [18F]F-AraG

INTERVENTIONS:
Drug: [18F]F-AraG

SUMMARY:
The goal of this study is to visualize biodistribution of a PET tracer called [18F]F-AraG through time in healthy human volunteers.

DETAILED DESCRIPTION:
A positron emission tomography (PET) imaging tracer will be intravenously injected into healthy human volunteers who provide informed consent. Following injection of this tracer each volunteer will have four whole-body PET scans inside a PET scanner to obtain images of tracer biodistribution at four different time points. This will allow studying the kinetics of the tracer as well analysis of tracer dosimetry. Safety of the tracer will also be analyzed in each volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects without history of chronic disease or at present an acute disease will be included.
* Ability to abide by the study conditions is also a requirement for inclusion.

Exclusion Criteria:

* Individuals under the age of 18 years and pregnant women will be excluded from the [18F]F-AraG imaging studies.
* Women who are breast-feeding will be excluded from the study.
* Individuals unable to provide informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Visualize biodistribution of the PET tracer [18F]F-AraG | 1 day
  Whole-body [18F]F-AraG PET scans will be performed at 4 different time points following intravenous injection of the PET tracer. Four whole-body images will be obtained that will reveal biodistribution of [18F]F-AraG at 4 different consecutive time points after intravenous injection.
Analyze human dosimetry of [18F]F-AraG | 1 day
  Time-Activity curves will be graphed by measuring activity in various organs at the 4 time points after tracer injection. From these time activity curves absorbed radiation will be calculated.
Assess acute safety of intravenously injected trace dose of [18F]F-AraG | 8 days
  Blood and urine samples may be collected at baseline and at 1 and 8 days after injection of [18F]F-AraG to perform metabolic panel, CBC and urine analysis. Vital signs and EKG will be measured and recorded at baseline, within 3 hours after tracer injection and at 1 and 8 days after tracer injection.

CONTACTS AND LOCATIONS:
Overall Officials: Henry VanBrocklin, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Imaging Center at China Basin, San Francisco, California, United States

REFERENCES:
- [Result] Namavari M, Chang YF, Kusler B, Yaghoubi S, Mitchell BS, Gambhir SS. Synthesis of 2'-deoxy-2'-[18F]fluoro-9-beta-D-arabinofuranosylguanine: a novel agent for imaging T-cell activation with PET. Mol Imaging Biol. 2011 Oct;13(5):812-8. doi: 10.1007/s11307-010-0414-x. PMID 20838911
- See also: Related Info — http://www.cellsighttech.com